CLINICAL TRIAL: NCT03313466
Title: Trial of Internet-Based Cognitive Behavioral Therapy for Insomnia in Patients Prescribed Insomnia Medications
Brief Title: Trial of Internet-Based Cognitive Behavioral Therapy for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Big Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11262
Record Dates: First submitted 2017-10-09; First posted 2017-10-18 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Artifacts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCBTI (Experimental): Intervention: An internet-based cognitive behavioral therapy program for insomnia (iCBTI) that is tailored to the individual's needs based on responses to questions.
  Interventions: Behavioral: Internet cognitive behavioral therapy for insomnia (iCBTI)
- Usual care (Active Comparator): Intervention: A group class on insomnia provided at each Kaiser Permanente Southern California medical center.
  Interventions: Behavioral: Class in sleeping well and improving insomnia

INTERVENTIONS:
Behavioral: Internet cognitive behavioral therapy for insomnia (iCBTI) — An internet-based program for providing individually tailored CBTI based on participant responses to questions and performance on weekly guided sleep strategies.
  Arms: iCBTI
Behavioral: Class in sleeping well and improving insomnia — A group education session providing advice on healthy sleep habits and ways to improve common forms of insomnia.
  Arms: Usual care

SUMMARY:
The investigators will conduct a randomized, controlled trial of internet-based cognitive behavioral therapy (iCBT) vs usual care for insomnia. The target population is patients prescribed medications for insomnia who have not had a dispensation of these medications in the preceding six months. The primary outcomes is dispensed days supply over the subsequent one year. Secondary outcomes include all types of health system clinical encounters. The investigators hypothesize that the group randomized into iCBT will have less insomnia medications dispensed than usual care controls, and less clinical encounters..

ELIGIBILITY:
Inclusion Criteria:

* A prescription for any of a set of selected insomnia medications.
* Age >18 years at the time of the prescription.
* A recent (<30 days before the prescription date) diagnosis of insomnia as determined by a set of selected International Classification of Disease (ICD) codes, to be used for medications that are not prescribed just for insomnia.
* Membership for >365 days prior to the prescription date.
* No evidence of a dispensed insomnia medication within six months (183 days) of the current prescription.

Exclusion Criteria:

* Contained in inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136630 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Days supply of dispensed insomnia medications | One year
  Days supply of dispensed insomnia medications up to one year after randomization.

SECONDARY OUTCOMES:
Health care inpatient and outpatient encounters | One year
  Number of physician or mid-level provider encounters (face-to-face, telephone, video): (1) outpatient, (2) acute care: emergency, inpatient, up to one year after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Derose, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Southern California, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derose SF, Rozema E, Chen A, Shen E, Hwang D, Manthena P. A population health approach to insomnia using internet-based cognitive behavioral therapy for insomnia. J Clin Sleep Med. 2021 Aug 1;17(8):1675-1684. doi: 10.5664/jcsm.9280. PMID 33908343